CLINICAL TRIAL: NCT02166281
Title: Impact of Adjuvant Treatment With Aromatase Inhibitor on Sleep Disturbances in Postmenopausal Women With Endocrine Responsive Early Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Study coordinators, Dr Rebecca Pedersini, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: Comfort
Record Dates: First submitted 2014-05-20; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Endocrine Responsive Early Breast Cancer
Keywords: Insomnia; Anxiety; Depression; Restless leg syndrome; Aromatase inhibitor; Body composition
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression; Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Insomnia is common in Breast cancer patients during adjuvant therapy with aromatase inhibitor.

However it is difficult to establish whether it is due to the knowledge of the disease or the treatment administred.

The investigators designed a cohort study in which questionnaires for the assessment of sleep quality (Pittsburgh Sleep Quality Index and Insomnia Severity Index), anxiety (State and Trait Anxiety Inventory), depression (Beck Depression Inventory), for the quality of life in general (Functional Assessment of Cancer Therapy) and for the evaluation of RLS (Restless Legs Syndrome Rating Scale) will be prospectively administered to patients with early breast cancer at baseline and during adjuvant treatment with aromatase inhibitors.

As secondary aims the investigators will also evaluate dietary and lifes' factors, born turn over and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Women with a histological diagnosis of invasive operated breast cancer (any pT, any pN)
* Women with more than 60 years
* Women less than 60 years with amenorrhea for at least 12 months and FSH and estradiol values in the range of menopause
* Signature of written informed consent.

Exclusion Criteria:

* Locally advanced or metastatic disease (M1)
* A history of breast cancer or other cancers diagnosed in the last 10 years, to exception of basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of severe osteoporosis before the diagnosis of breast cancer
* Bisphosphonate therapy before the diagnosis of breast cancer
* Other serious medical conditions that could limit the ability of the patient to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal Women with early stage endocrine responsive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
The number of participants who suffer from insomnia | 24 months
  We use some validated questionnaires to measure this item

SECONDARY OUTCOMES:
The number of participants who suffer from anxiety and depression | 24 months
  We use some validated questionnaires to measure this item
The number of participants who suffer from Restless | 24 months
  We use some validated questionnaires to measure this item
Correlating the onset of restless with anxiety, depression and insomnia | 24 months
  We analyse correlation into the database
Describe changes in lean body mass, fat mass, bone mineral density during treatment | 24 months
  We analyse this items after DEXA
The number of participants with abnormal level of vitamin d | 24 months
  We asses participants with levels of vitamin out of range
Correlate the changes in body composition with circulating levels of vitamin D | 24 months
  We use statistic software to asses changes
Number of fracture and their correlation with the density bone mineral and other parameters of body composition | 24 months
  We use statistic software to asses correlation

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca RP Rebecca, Pedersini, Principal Investigator — Azienda Spedali Civili Brescia
Locations (1):
- Azienda Spedali Civili Brescia DH Oncologia, Brescia, Brescia, Italy

REFERENCES:
- [Background] 1.Early Breast Cancer Trialists' Collaborative Group.Lancet 2005;365:1687-1717. 2.Slamon D, Eiermann W, Robert N, et al. NEJM 2011;365:1273-1283. 3.The Arimidex, Tamoxifen, Alone or in Combination (ATAC) Trialists' Group, et al. Lancet Oncol, 2008;9:45-53. 4. The BIG 1-98 Collaborative Group. New Engl J Med 2009;361:766-776. 5. Dowsett M, Cuzick J, Ingle J, et al. J Clin Oncol 2010;28:509-518. 6. Forbes JF, Cuzick J, Buzdar A et al. Lancet Oncol 9: 45-53, 2008 7. Monnier A. Eur J Cancer Supplements 2008;6 (7):113. 8.Bower JE. J Clin Oncol. 2008, 10;26(5):768-77. 9. Desai K, Mao JJ, Su I, Demichele A, Li Q, Xie SX, Gehrman PR. Support Care Cancer. 21(1):43-51, 2013 10. Lockefeer JPM, De Vries J. Psico-oncology 2013;22(5):1127-33 11. Julienne E. Bower, Patricia A. Ganz, Michael R. Irwin, et al.J Clin Oncol. 2011,29;26(10):3517-3522. 12. Floortje Mols A, Vingerhoets B, Jan Willem Coebergh A. European Journal of Cancer 41: 2613-2619, 2005 13.Meunier A, Bachelot T, leynet E, et al. San Antonio Breast Cancer Symposium, 2008 14 Saini A, Berruti A, Ferini-Strambi L, et al. Pain Symptom Manage. 2013;46(1):56-64. 15. Luca Ostacoli, Andrea Saini, Luigi Ferini-Strambi et al. Qual Life Res, 2010 16 Tredan O, Bajard A, Meunier A, et al.Clin Nutr 29(2):187-191, 2010; 17. Harvie MN, Campbell IT, Baildam A, et al. Breast Cancer Res Treat 83(3):201-210, 2007 18. Goodwin PJ, Ennis M, Pritchard KI, et al. J Clin Oncol 17(1):120-129, 1999 19.Hoskin PJ, Ashley S, Yarnold JR. Breast Cancer Res Treat 22(2):129-132, 1992 20.Camoriano JK, Loprinzi CL, Ingle JN, Therneau TM, Krook JE,Veeder MH (1990) J Clin Oncol 8(8):1327-1334,
- [Background] 21. Chlebowski RT, Weiner JM, Reynolds R, Luce J, Bulcavage L, Bateman JR (1986) Breast Cancer Res Treat 7(1):23-30) 22 Demark-Wahnefried W, Winer EP, Rimer BK (1993) J Clin Oncol 11(7):1418-1429). 23 Demark-Wahnefried W, Hars V, Conaway MR, et al. Am J Clin Nutr. 1997;65(5):1495-501 24 Demark-Wahnefried W, Rimer BK, Winer EP (1997) J Am Dietetic Assoc, 97(5):519-526, 529 (quiz 527-518) 25.Fisher B, Dignam J, Bryant J, et al. J Natl Cancer Inst 88(21):1529-1542, 1996 26. Day R, Ganz PA, Costantino JP, et al. J Clin Oncol 17(9):2659-2669, 1999 27. Powles T, Eeles R, Ashley S, et al. Lancet 352(9122):98-101 , 1998 28 Wahnefried WD, Campbell KL, Hayes SC. Cancer 15: 2277- 2287, 2012 29. Van Londen GJ, Perera S, Vujevich K, et al. Breast Cancer Res Treat; 125(2): 441-446, 2011 30 Berrino F, Pasanisi P, Bellati C I nt J Cancer 113: 499-502, 2005 31.Goodwin PJ, Ennis M, Pritchard KI, et al. J Clin Oncol. 2012 Jan 10;30(2):164-71. 32. Duggan C, Irwin ML, Xiao L, et al. J Clin Oncol. 2011 Jan 1;29(1):32-9. 33 Rabaglio M, Sun Z, Prince KN, et al. Ann Oncol 20: 1489-1498, 2009 34 Hillner BE, Ingle JN, Chlebowski RT, et al. J Clin Oncol. 2003 1;21(21):4042-57. 35.Kanis J, Borgstrom F, De Laet C, et al. Int 16: 581-589; 2005 36. Berruti A, Tucci M, Mosca A, Vana F et al. J Clin Oncol., 10;25(11):1455-6, 2007 37 Bischoff-Ferrari HA, Giovannucci E, Willet WC, et al. Am J clin Nutr 2006; 84: 18 38 Rastelli AL, Taylor ME, Gao F, et al. Breast Cancer Res Treat, 2011 107-16, 2011 39. Singh S, Cuzick J, Mesher D, et al. Breast cancer Res Treat 2012: 132: 625-629 40. Helzlsouer KJ, Gallicchio L, MacDonald R, et al. Breast Cancer Res Treat 2012; 131 (1): 277-85
- [Background] 41 Park S, Ham JO, Lee BK. Clin Nutr, 2013 S0261-5614(13)00256-2. 42 Buttigliero C, Monagheddu C, Petroni P, et al. Oncologist.16(9):1215-27, 2011 43 Otte J, Rand K, carpenter J et al. Journal of pain and symptom management: 1-8; 2012 44 Buysse DJ, Reynolds CF, Monk TH, et al. Psychiatry res 28: 193-213, 1989 45 Zigmond AS, Snaith RP. Acta psychiatr scand 1983; 67: 361-370 46 Brady MJ, Cella DF, Mo F. J Clin Oncol 15; 974-986, 1997 47 Abetz L, Arbuckle R, Allen RP, et al. Sleep Med 2006;7:340-349. 48.Coombes RC, Kilburn LS, Snowdon CF et al. Lancet 369: 559-570, 2007 49 Linee guida Rete oncologica lombarda 50. Hillner BE, Ingle JN, Chlebowski RT, et alClin Oncol 21:4042-4057, 2003 51. Gralow JR, Biermann JS, Farooki A, et al. J Natl Compr Canc Netw 7:S1-S32, 2009; S33-S35 (suppl 3) 52. Hadji P, Aapro MS, Body JJ, et al. Ann Oncol 22:2546-2555, 2011 53. Rizzoli R, Body JJ, De Censi A, et al. Osteoporos Int [epub ahead of print on January 20, 2012] 54. Body JJ, Bergmann P, Boonen S, et al. Osteoporos Int 18:1439-1450, 2007 55.David M, Julie D, , Richard E, et al. A consensus position statement from a UK Expert Group Cancer Treatment Reviews (2008) 34, S3- S18 56.Savard MH, Savard J, Simard S et al. Psycho-Oncology 14:429-441, 2005 57. Spielberger C. Consulting Psychologists Press; 1983. 58. Beck AT, Ward CH, Mendelson M, Mock J, Erbaugh J. Arch Gen Psychiatry. 1961 Jun;4:561-71. 59. Lichstein KL, Stone KC, Donaldson J et al. Sleep 29(2): 232-239, 2006. 60.Sack RL, Pires ML, Brandes RW et al.Vol. 24 Supplement Abstract #719.R, pg.A405, Sleep 2001. 61. King MA, Jaffre MO, Morrish E et al. Sleep Medicine 6(4): 1-7, 2005.